CLINICAL TRIAL: NCT06174662
Title: The Effect of Music on Procedural Distress During Mobilization in Intensive Care Unit Patients: A Randomized Controlled Trial
Acronym: MUSICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Filip Haegdorens, Assistant professor, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MUSICU
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Pain; Stress; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT) with parallel arms: control and intervention group. Not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): Music through noise cancelling headphones.
  Interventions: Device: Music
- No music (No Intervention): Control group receiving regular care. No music will be offered to the patient.

INTERVENTIONS:
Device: Music — The patient can decide the music genre (a standard playlist) and receives a noise-cancelling headphone playing the chosen music during mobilization.
  Arms: Music

SUMMARY:
This intervention study will investigate the effects of music therapy on procedural distress, the overall experience of pain, anxiety, and stress, during the procedure of sitting up in a chair for patients admitted to the intensive care unit (ICU).

DETAILED DESCRIPTION:
There is a paucity of literature on the use of music therapy ('music care') in intensive care units (ICUs) during the process of mobilization. However, research suggests that mobilization can reduce the risk of depression and improve cognitive function (Chiang et al., 2006). This study aims to investigate the impact of music therapy on procedural comfort during sit-to-stand mobilization in ICU patients.

Specifically, the investigators seek to examine the effects of music therapy on pain perception, stress levels, anxiety levels, and vital parameters (blood pressure, heart rate, and respiratory rate) during this procedure. The investigators hypothesize that music therapy can improve procedural comfort by reducing pain, stress, and anxiety.

This study employs quantitative multicenter research, specifically a randomized controlled trial (RCT), involving ICU patients at three hospitals: AZ Monica Deurne, GZA campus Sint-Augustinus, and Sint-Vincentius.

During the intervention, patients will listen to their preferred music through noise-canceling headphones. Patients will be able to select their preferred music.

To assess the effects of music therapy, the investigators developed a self-designed measurement tool, validated using content validation indices (CVI) with an expert panel including pain nurses. The tool measures various indicators, including:

Vital parameters: (arterial) blood pressure, heart rate, and respiratory rate

Pain perception: Using an 11-point Likert scale from 0 to 10, nurses will assess the patient's pain level. Zero indicates no pain, while 10 represents the worst imaginable pain.

Anxiety and stress levels: Nurses will utilize 11-point Likert scales from 0 to 10 to measure the patient's anxiety and stress levels. The sum of these three scores will provide an overall measure of procedural distress.

To assess the duration of the effects of music therapy, we will record the above indicators at four time points:

Time 0: Ten minutes before sit-to-stand mobilization begins

Time 1: Ten minutes after sit-to-stand mobilization is completed

Time 2: Immediately before returning the patient to bed, after music stops

Time 3: Ten minutes after the patient is back in bed

Delta calculations will be performed to measure changes between time points.

The selected music playlist will be briefly noted on the measurement tool, and a final Likert scale will assess patient satisfaction with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* They are admitted to the ICU
* They have a Richmond Agitation-Sedation Scale (RASS) score of +1, 0, or -1
* They are able to speak Dutch

Exclusion Criteria:

* They are younger than 18 years old
* They have a hearing impairment
* They are in isolation
* They have a cranial dressing or intracranial pressure monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
pain perception level | Ten minutes before mobilization begins and ten minutes after mobilization is completed
  Using an 11-point Likert scale from 0 to 10, nurses will assess the patient's pain level
stress perception level | Ten minutes before mobilization begins and ten minutes after mobilization is completed
  Using an 11-point Likert scale from 0 to 10, nurses will assess the patient's stress level.
anxiety perception level | Ten minutes before mobilization begins and ten minutes after mobilization is completed
  Using an 11-point Likert scale from 0 to 10, nurses will assess the patient's anxiety level.

SECONDARY OUTCOMES:
Time of mobilization | Ten minutes before mobilization begins and ten minutes after mobilization is completed
  Time in minutes of mobilization
Blood pressure | Ten minutes before mobilization begins and ten minutes after mobilization is completed
  Systolic Blood Pressure
Heart rate | Ten minutes before mobilization begins and ten minutes after mobilization is completed
  Heart frequency per minute
Respiratory frequency | Ten minutes before mobilization begins and ten minutes after mobilization is completed
  Respiratory frequency per minute

CONTACTS AND LOCATIONS:
Locations (1):
- University of Antwerp, Wilrijk, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared on request